CLINICAL TRIAL: NCT01784237
Title: Comparison Between an Anterior Rhinoscopic Scoring Scale With the Sniff Test to Predict Nasal Insertability Before Transnasal Endoscopy: A Prospective, Randomized, Controlled Study
Brief Title: A Novel Anterior Rhinoscopic Scoring Scale to Predict Nasal Insertability Before Transnasal Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Chi-Tan Hu, Chief, Division of Gastroenterology, Buddhist Tzu Chi General Hospital, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB101-77
Record Dates: First submitted 2012-12-12; First posted 2013-02-05 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Injury Due to Endoscopic Examination; Transnasal Endoscopy Induced Epistaxis; Transnasal Endoscopy Induced Nasal Pain
Keywords: Endoscopes; Esophago-gastro-duodenoscopy; Transnasal endoscopy; Anterior meatoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anterior meatuscopy (Experimental): All patients in the study group receive anterior meatoscopy whereas patients in the control group perform a sniff test to select the most patent nostril for nasal anesthesia and transnasal endoscopic insertion.
  Interventions: Procedure: anterior meatoscopy
- Nasal sniff test (Active Comparator): A sniff test for nasal patency is a common method before ultrathin transnasal esophago-gastro-duodenoscopy (UT-EGD) to select the right or left nostril for insertion.
  Interventions: Procedure: Nasal sniff test

INTERVENTIONS:
Procedure: anterior meatoscopy — The nasal vestibule is the most anterior part of the nasal cavity. It is lined by the same epithelium of the skin (stratified squamous epithelium) but not respiratory epithelium (pseudostratified columnar ciliated epithelium) so that an endoscope tip in this region would hardly causes trauma or bleeding. Before being inserted gently into the nasal vestibule for anterior rhinoscopy, the endoscope tip is applied with 2% lidocaine gel and then sprayed with 10% liquid lidocaine. This procedure can provide mild vestibular anesthesia which can prevent patients from sneezing when the vibrissae hair is irritated by the endoscope tip. Instead of holding the insertion tube as usual, an endoscopist holds the bending section for better control of the distal tip during anterior meatuscopy.
  Arms: Anterior meatuscopy
Procedure: Nasal sniff test — All patients in the control group receive a sniff test in the left lateral decubitus (LLD) position directed and recorded by an assistant nurse. This test has been conducted for decades and is still used by many transnasal endoscopists, otolaryngologists, and pediatrics. In brief, the more patent nostril is selected by the patient inhaling through only one nostril with the other sealed by the examiner's index ﬁnger. Patients are asked to indicate which of their nostrils is most patent. If neither is more patent, the right nostril is chosen by default. The middle meatus is more difficult to examine and may be less well anesthetized than other structures. Thus, the inferior nasal meatus is selected for each case because the inferior meatus is usually the largest of the three nasal meatuses.
  Arms: Nasal sniff test

SUMMARY:
A sniff test for nasal patency is a common method before ultrathin transnasal esophago-gastro-duodenoscopy (UT-EGD) to select the right or left nostril for insertion, yet there is no objective method to select an appropriate meatus insertion site (MIS) where tolerance and epistaxis rate can be improved.

The investigators hypothesize that that an objective anterior rhinoscopy (to be more specific, the investigators term it "anterior meatoscopy") method might be more effective than the subjective breathing-in method (sniff test) to select the appropriate meatus insertion site, thus reducing nasal bleeding and nasal discomfort.

The aim of this study is to evaluate the effectiveness of an endoscopic meatus scoring scale (EMSS) by anterior meatoscopy (AM) to select a MIS on patient tolerance and adverse events during nasal anesthesia and UT-EGD.

The investigators will perform a prospective randomized-controlled trial to compare patient tolerability and adverse events during nasal anesthesia and endoscopy between the AM-selected and self-selected MIS. A total of 233 consecutive patients with epigastric discomfort (symptoms of non-ulcer dyspepsia) will be included in the study in a large tertiary referral hospital in Taiwan.

DETAILED DESCRIPTION:
Transnasal esophago-gastro-duodenoscopy (UT-EGD) offers physicians and patients a number of advantages compared with conventional peroral EGD (P-EGD) and has become increasingly popular in clinical practice over the past several years. However, insertion failure varying from 2.3% to 62.7% due to tight nasal vault have been reported. Dumortire reported 17.9 % of patient refused UT-EGD due to nasal pain and epistaxis remains to be a common side effect. Therefore a well performed nasal anesthesia has been regarded as the most important step for UT-EGD.

The concept of endoscopic guidance is actually an application of anterior rhinoscopy to select the most patent meatus for nasal anesthesia and endoscopic insertion. The scope should be placed in the side of the nasal cavity that is most patent. Therefore, it is reasonable that a nasal examination is performed prior to UT-EGD to determine the less obstructed side.

In fact, anterior rhinoscopy is a common outpatient procedure by otolaryngologists and is performed with an otoscope. Instead, we use a transnasal endoscope to select the most patent meatus and thus we first introduce the concept of anterior "meatus-copy", which is different from "meatoscopy" for the urinary meatus.

The conventional sniff nasal patency test is an inspection of nasal passability by asking a patient to compare the breathing-in air flow in either side of the nose. This is a self-selected and subjective method of choosing just the right or left nostril for transnasal endoscopy.

Nasal septum and nasal turbinates, especially the inferior turbinates, are erectile tissues in the nose, fluctuate greatly in size depending on physiological changes (e.g. body temperature and exercise) and response to inflammation. Often, the sensation of a blocked nose is subjective. The otolaryngologist may find a perfectly patent airway and yet the patient will insist that his nose is clogged up. Therefore, an objective method to evaluate nasal patency would help to avoid a narrowed meatus, thereby reducing nasal pain and epistaxis during nasal anesthesia and transnasal endoscopy.

Methods used to objectively measure nasal patency and resistance include rhinomanometry and acoustic rhinometry. However, these two methods are sophisticated and not straightforward. There is no literature describing the optimal selection method for transnasal endoscopic insertion. Assessments of nasal patency by dynamic methods include nasal peak flow, rhinomanometry, and acoustic rhinometry. However, a convenient endoscopic method of evaluating nasal meatus patency has not been proposed.

Locating on the anterior portion of a meatus, the transnasal endoscope itself can act as a nasoscope to look for the most patent meatus.

We found anterior meatuscopy allows the direct visualisation of the turbinates and meatus without causing discomfort. Thus it may be a useful ancillary technique to select the most patent meatus for scope insertion. Hence, the primary objective of this study is to evaluate whether a anterior meatuscopy scoring system could reduce nasal bleeding and improve tolerance associated with UT-EGD.

ELIGIBILITY:
Inclusion Criteria:

All outpatients with epigastric discomfort (non-ulcer dyspepsia), aged 18-65 years are eligible for this study.

Exclusion Criteria:

Patients who have prior nasal trauma or surgery, recent or present upper gastrointestinal bleeding and coagulopathy are excluded from this study. Patients who are allergic to an anesthetic agent and who have uncontrolled hypertension or coronary artery disease are not recruited. Those who are uncooperative and unable to answer questions are also excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measures were tolerability proﬁles on a validated visual analogue scale | Immediately after transnasal endoscopy up to all questionnaires answered (about 15 minutes)
  The primary outcome measures were tolerability proﬁles on a validated visual analogue scale as previously described and difficulty in inserting the transnasal endoscope through the selected meatus based on a Likert scale. The scale contained 5 points of difficulty: minimal, slight, moderate, substantial, and extreme. Facing a 5-point VAS card (1 = minimal discomfort to 5 = severe discomfort), all patients gave realtime feedback by speaking or pointing out their scorings for the following: (1) pain during anesthesia, (2) pain during nasal insertions, and (3) pain during exsertion, and they answered immediately after UT-EGD for (4) overall tolerance.

SECONDARY OUTCOMES:
Secondary outcome measure evaluates the side effects of transnasal endoscopy | Immediately after transnasal endoscopy up to all questionnaires answered (about 15 minutes)
  Secondary outcome measures were evaluated by assisting nurses, who recorded epistaxis, patient's willingness to receive the same procedure the next time, and post-procedural side effects including headache, light headiness, mucous discharge, and confirmed sinusitis by otolaryngologist. The visual capacity for the anterior nasal cavity ranking on a 5-point scale (5 represented standard EGD and 1 poor visual quality) was as previously described

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Tan Hu, MD, PhD, Principal Investigator — Budhist Tzu Chi Hospital and Tzu Chi University
Locations (1):
- Buddhist Tzu Chi Hospital, Hualien City, Hualien county, Taiwan